CLINICAL TRIAL: NCT07127757
Title: Clinical Evaluation of Visual Outcomes With the Wavelight Plus Excimer Laser in Normal and Dim Lighting
Brief Title: Clinical Evaluation of WaveLight Plus LASIK
Status: Recruiting | Type: Observational
Sponsor: Laser Defined Vision (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: KS-25-01
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Wavelight Plus LASIK
  Interventions: Device: Wavelight Plus LASIK

INTERVENTIONS:
Device: Wavelight Plus LASIK — Wavelight plus LASIK is an advanced laser eye surgery technology designed to enhance visual outcomes through personalized treatment plans. This system integrates comprehensive diagnostics, including biometry, tomography, and wavefront measurements, to create a tailored ablation profile for each patient.

SUMMARY:
This study is a single-site, single-arm, prospective, observational study of subject satisfaction, quality of vision, and quality of life after bilateral LASIK surgery. Subjects will be assessed up to 3 months post-operatively. Clinical evaluations will include refractive outcomes, visual acuity, and administration of the adapted PROWL and Low Luminance Questionnaire (LLQ-32) Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to understand and sign an IRB approved Informed consent form
* Willing and able to attend all scheduled study visits as required per protocol
* Minimum of 18 years of age
* Myopia up to -8.00 D, astigmatism up to -3.00 D, with SE more than -1.00D and up to -9.00D, based on Sightmap measured refraction
* Best corrected photopic distance visual acuity of 20/20-2 or better (≤ 0.04 logMAR)
* Mesopic pupil size ≥ 4.5mm
* Less than 0.75 D manifest refraction spherical equivalent difference between Sightmap refraction and subjective manifest refraction
* Stable refraction (within ± 0.50 D) as determined by manifest refraction spherical equivalent for a minimum of 12 months prior to surgery, verified by consecutive subjective refractions or medical records or prescription history
* If currently wearing contact lenses:

  * Soft CTL wearers discontinue for minimum 3 days prior to first refraction
  * RGP or toric soft CTL wearers discontinue for ≥2 weeks prior to first refraction

Exclusion Criteria:

* Subjects who are pregnant or nursing
* Acute or chronic disease or illness that would increase the operative risk or confound the outcomes of the study
* Patients with flap complications
* Systemic medications that may confound the outcome of the study or increase the risk to the subject.
* Ocular condition (other than high myopia) that may predispose the subject to future complications, such as ectasia
* History or evidence of active or inactive corneal disease (e.g., herpes simplex keratitis, herpes zoster keratitis, recurrent corneal erosion syndrome, corneal dystrophy)
* Evidence of retinal vascular disease
* Keratoconus or Keratoconus suspect
* Glaucoma or glaucoma suspect by exam findings and/or family history
* Previous intraocular or corneal surgery
* Predicted residual stromal bed thickness < 250 μm
* Intended to have monovision treatment
* Participation in other current clinical trials

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible test subjects will be 18+ years of age and who are candidates for Wavelight Plus LASIK to correct myopia or myopic astigmatism. Patients who are eligible for LASIK surgery with the Wavelight Plus device may undergo the procedure even if they choose not to participate in the research study. The decision to perform surgery with the device will be made based on clinical indications, irrespective of participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
% of eyes with UDVA of 20/10, 20/12.5, 20/16 and 20/20 in photopic conditions at 3 months (monocular and binocular) | 3 months postoperatively
% of eyes with UDVA of 20/10, 20/12.5, 20/16 and 20/20 in mesopic conditions at 3 months (monocular and binocular) | 3 months postoperatively
% of eyes with CDVA of 20/10, 20/12.5, 20/16 and 20/20 in photopic conditions at 3 months (monocular and binocular) | 3 months postoperatively

SECONDARY OUTCOMES:
% of eyes that achieve UDVA equal to or better than preoperative CDVA | 3 months postoperatively
% of eyes with lines gained/lost lines (post-up UDVA VS pre-op CDVA) | 3 months postoperatively
% of eyes with absolute MRSE within +/- 0.25, 0.50, 0.75, and 1.00D at 3 months | 3 months postoperatively
% of eyes that achieved manifest refraction cylinder within +/- 0.25, 0.50, 0.75, and 1.00D at 3 months | 3 months postoperatively
Patient-Reported Outcomes with the modified PROWL Questionnaire and Low Luminance Questionnaire (LLQ-32) at 3 months | 3 months postoperatively

OTHER OUTCOMES:
% of eyes with 10% contrast UDVA (mesopic, binocular) of 20/10, 20/12.5, 20/16, 20/20 and 20/25 at 3 months | 3 months postoperatively
% of eyes with 10% contrast CDVA (mesopic, binocular) of 20/10, 20/12.5, 20/16, 20/20 and 20/25 at baseline and 3 months | 3 months postoperatively
% of eyes with UDVA of 20/8 in photopic conditions at 3 months (monocular and binocular) | 3 months postoperatively
% of eyes with CDVA of 20/8 in photopic conditions at 3 months (monocular and binocular) | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Karl Stonecipher, MD, Principal Investigator — Laser Defined Vision
Locations (1):
- Laser Defined Vision, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No